CLINICAL TRIAL: NCT00249067
Title: The Retrospective Evaluation of Carvedilol Versus Captopril and Digoxin/Lasix Therapy in Congestive Heart Failure Due to Left-to-Right Shunt Lesions
Brief Title: Retrospective Evaluation of Carvedilol Versus Captopril in CHF Patients
Status: Terminated | Type: Observational
Why Stopped: data collection completed
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05.178
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Heart Failure; Heart Murmurs
Keywords: Congestive Heart Failure, Left-to-Right Shunt
MeSH Terms: conditions — Heart Failure; Heart Murmurs

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review examining our experience with carvedilol in CHF secondary to left-to-right heart shunt lesions. The treatment group will be children who have received carvedilol. The control or comparison groups will be patients who have received either digoxin/furosemide or captopril for this indication. Charts will be reviewed of patients who have been treated at Children's Healthcare of Atlanta and as outpatients by Sibley Heart Center Cardiology between September 2000 and October 2005. Patients will have been started on carvedilol prior to April 1, 2005 and only information up to October 1, 2005 will be used for this study. We will review approximately 50 charts for this study.

We will evaluate the effectiveness of these medications at reducing symptoms of CHF.

DETAILED DESCRIPTION:
This is a retrospective chart review examining our experience with carvedilol in CHF secondary to left-to-right heart shunt lesions. The treatment group will be children who have received carvedilol. The control or comparison groups will be patients who have received either digoxin/furosemide or captopril for this indication. Charts will be reviewed of patients who have been treated at Children's Healthcare of Atlanta and as outpatients by Sibley Heart Center Cardiology between September 2000 and October 2005. Patients will have been started on carvedilol prior to April 1, 2005 and only information up to October 1, 2005 will be used for this study. We will review approximately 50 charts for this study.

We will evaluate the effectiveness of these medications at reducing symptoms of CHF.

ELIGIBILITY:
Inclusion Criteria: Children aged 0-18 years with a cardiac defect resulting in a left-to-right shunt (i.e. ventricular septal defect) who develop congestive heart failure. Patient must have been treated with one of the study medications: carvedilol, digoxin, or furosemide.

-

Exclusion Criteria: Patients who are not between 0-18, who do not have a defect resulting in left-to-right shunt, who do not have congestive heart failure and who have not been treated with one of the study medications: carvedilol, digoxin, or furosemide.

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2005-10; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Dayton, MD, Principal Investigator — Resident-Emory Department of Pediatrics
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States